CLINICAL TRIAL: NCT00708279
Title: Study of Osteopathic Manipulation in the Management of Angina
Acronym: SOMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: Osteopathic Heritage Foundations (Other)
Responsible Party: Joy L. Palmer, D.O., Principal investigator, Edward Via College of Osteopathic Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-07-04 SOMMA; F-07-04 AOA/OHF Fellowship (Other: American Osteopathic Association - Osteopathic Heritage Fund)
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-06

CONDITIONS: Angina Pectoris
Keywords: angina pectoris, osteopathic manipulation
MeSH Terms: conditions — Angina Pectoris | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): After establishing a baseline for the first 4 weeks of trial involvement, thereby providing their own control group, all participants begin the intervention phase of osteopathic manipulation.
  Interventions: Procedure: Osteopathic manipulation

INTERVENTIONS:
Procedure: Osteopathic manipulation — Participant will be evaluated and treated for somatic dysfunction utilizing osteopathic manipulation once a week for 3 weeks, then once every 3 weeks for three more visits; a total of 6 interventions in 3 months.
  Other Names: osteopathic manipulative medicine; structural exam; viscero-somatic reflexes; circulatory-respirtatory model; musculoskeletal model

SUMMARY:
The purpose of this study is to assess the effectiveness of osteopathic manipulation in decreasing angina pectoris symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Canadian Cardiovascular Society Class II, III for a minimum of 6 months
* documented coronary artery disease via previous myocardial infarction, abnormal stress test, or abnormal coronary angiogram of greater than or equal to 50% luminal obstruction of at least one epicardial vessel.

Exclusion Criteria:

* severe left ventricular dysfunction
* symptomatic heart failure
* symptomatic aortic stenosis or any valvular disease
* significant pulmonary disease
* unstable angina
* major surgery or angioplasty in the past three months
* acute myocardial infarction within past three months
* insulin dependent diabetes mellitus
* uncontrolled hypertension
* acute renal or hepatic failure
* currently being treated with osteopathic manipulation

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Decrease in angina symptoms | over 4 month period

SECONDARY OUTCOMES:
Improvement in quality of life | over 4 month period

CONTACTS AND LOCATIONS:
Overall Officials: Joy L. Palmer, D.O., Principal Investigator — University of New England
Locations (1):
- University Health Care, Saco, Maine, United States